CLINICAL TRIAL: NCT06051617
Title: AFFIRM: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Seladelpar on Clinical Outcomes in Patients With Primary Biliary Cholangitis (PBC) and Compensated Cirrhosis
Brief Title: Seladelpar in Subjects With Primary Biliary Cholangitis (PBC) and Compensated Cirrhosis
Acronym: AFFIRM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB8025-41837; 2024-516525-31-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis (PBC); PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — seladelpar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seladelpar (Experimental)
  Interventions: Drug: Seladelpar
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seladelpar — * Seladelpar 10 mg one capsule daily for up to 36 months in participants with CP-A cirrhosis or
  * Seladelpar 5 mg one capsule daily for up to 36 months in participants with CP-B cirrhosis.
  Other Names: Livdelzi®
  Arms: Seladelpar
Drug: Placebo — One capsule daily for up to 36 months.
  Arms: Placebo

SUMMARY:
To Evaluate the Effect of Seladelpar on Clinical Outcomes in Patients with Primary Biliary Cholangitis (PBC) and Compensated Cirrhosis.

DETAILED DESCRIPTION:
To Evaluate the Effect of Seladelpar on Clinical Outcomes in Patients with Primary Biliary Cholangitis (PBC) and Compensated Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet the following criteria to be eligible for study participation:

1. Must be at least 18 years old.
2. Must have a confirmed prior diagnosis of PBC
3. Evidence of cirrhosis
4. CP Score A or B
5. Females of reproductive potential must use at least 1 barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male individuals who are sexually active with female partners of reproductive potential must use barrier contraception, and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose
6. Individuals must be able to comply with the instructions for study drug administration and be able to complete the study schedule of assessments (SOA)

Exclusion Criteria:

Individuals must not meet any of the following criteria to be eligible for study participation:

1. Prior exposure to seladelpar
2. A medical condition other than PBC that, in the Investigator's opinion, would preclude full participation in the study
3. History of liver transplantation or actively listed for cadaveric or planned living donor transplant.
4. Decompensated cirrhosis
5. Evidence of portal vein thrombosis based on imaging at time of Screening by Doppler ultrasound or prior evidence by CT or MRI
6. Hospitalization for liver-related complication within 12 weeks of Screening
7. Laboratory parameters at Screening:

   1. Alkaline phosphatase (ALP) < 1.5× Upper limit of normal (ULN) or ≥ 10×ULN
   2. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≥5×ULN
   3. Total bilirubin (TB) ≥5×ULN
   4. Platelet count ≤50×10^3/µL
   5. Albumin ≤2.8 g/dL
   6. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m^2
   7. MELD score >12. For individuals on anticoagulation medication, baseline International normalized ratio (INR) determination for MELD score calculation should take anticoagulant use into account, in consultation with the Medical Monitor.
   8. Serum alpha-fetoprotein (AFP) >20 ng/mL
   9. INR >1.7
8. CP-C cirrhosis
9. History or presence of other concomitant liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 36 months
  EFS as measured by the time from start of treatment to the first occurrence of any of the following clinical events:
  1. Death by any cause;
  2. Liver transplantation;
  3. MELD score ≥15;
  4. Ascites requiring treatment;
  5. Hospitalization for any of the following:
     1. Esophageal or gastric variceal bleeding
     2. Hepatic encephalopathy
     3. Spontaneous bacterial peritonitis

SECONDARY OUTCOMES:
Overall survival | 36 months
  Time from start of treatment to death from any cause.
Liver transplant-free survival | 36 months
  Time from start of treatment to the first occurrence of liver-related death or liver transplantation.
Time to hospitalization | 36 months
  Time from start of treatment to the first occurrence of hospitalization for qualifying PBC clinical events
Time to Event Free Survival (EFS) | 36 months
  1. MELD score ≥15
  2. Ascites requiring treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (159):
- United States (45):
  - St. Joseph's Hospital and Medical Center - 350 W. Thomas, Phoenix, Arizona
  - OM Research LLC, Lancaster, California
  - SCPMG/Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedar Sinai Medical Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Stanford University, Redwood City, California
  - University of California, Davis Medical Center, Sacramento, California
  - California Pacific Medical Center - Sutter Pacific Medical Foundation, San Francisco, California
  - Connie Frank Transplant Center at UCSF, San Francisco, California
  - Covenant Metabolic Specialists, LLC, Fort Myers, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - Florida Research Institute, Tampa, Florida
  - Piedmont Atlanta Hospital / Piedmont Transplant Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - University of Louisville, Clinical Trials Unit, Louisville, Kentucky
  - Ochsner Clinic Foundation, Jefferson, Louisiana
  - University Health System - East Jefferson General Hospital Campus, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Medical Center - Columbus, Detroit, Michigan
  - University of Rochester Medical Center - Strong Memorial Hospital, Rochester, Minnesota
  - Northwell Health Center for Liver Disease and Transplantation, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hosptials Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - Gastro One, Cordova, Tennessee
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Professional Office Building One, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
  - MedStar Health Research Institute / MedStar Georgetown Transplant Institute at Fairfax, Fairfax, Virginia
  - Maryview Hospital LLC d/b/a Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - VCU Health Clinical Research Services Unit (CRSU), Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Argentina (8):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Consultorios Médicos Dr. Doreski - PPDS, Buenos Aires
  - Buenos Aires Mácula, Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, Buenos Aires
  - AES - AS - Glenny Corp. S.A. Buenos Aires, Buenos Aires
  - Higea S.A., Mendoza
  - DIM Clinica Privada, Ramos Mejía
  - CINME S.A. - Centro de Investigaciones Metabólicas, Recoleta
- Australia (5):
  - Princess Alexandra Hospital, Queensland, Queensland
  - Flinders Medical Center, Adelaide, South Australia
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Northern Health, Epping, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Austria (4):
  - Landeskrankenhaus Hall, Hall in Tirol
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH - Standort Wels, Wels
- Belgium (2):
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
- Canada (6):
  - University of Calgary, Calgary
  - University of Alberta, Edmonton
  - Centre Hospitalier de l'Universite de Montreal, Montreal
  - Ottawa Hospital, Ottawa
  - Diex Recherche - Québec - PPDS, Québec
  - GI Research Institute Foundation, Vancouver
- Chile (4):
  - Centro de Investigación y Prevención Cardiovascular, La Serena
  - Pontificia Universidad Católica de Chile, Santiago
  - BIOCINETIC Ltda, Santiago
  - Clinical Research Chile SpA - PPDS, Valdivia
- China (13):
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Hospital of Nanjing, Nanjing
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang
  - Henan Provincial People's Hospital, Zhengzhou
  - The Third People's Hospital of Zhenjiang, Zhenjiang
- RESEARCH Site s.r.o, Pilsen, Czechia
- Aarhus Universitetshospital, Aarhus, Denmark
- France (6):
  - Hôpital Claude Huriez-Lille-1 Place de Verdun, Lille
  - Hospices Civils de Lyon (HCL) - Hopital de la Croix-Rousse, Lyon
  - CHU-Montpellier-Hopital St Eloi, Montipellier
  - Hopital Saint Antoine, Assistance Publique-Hopitaux de Paris, Paris
  - AP-HP Hopital Henri Mondor, Paris
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
- Germany (3):
  - Charité Campus Virchow-Klinikum-Augustenburger Platz 1, Berlin
  - Universitatsklinikum des Saarlandes, Homburg
  - Gastroenterologisch - Hepatologisches MVZ Kiel GmbH, Kiel
- Greece (3):
  - Evangelismos General Hospital, Athens
  - University General Hospital of Larissa, Larissa
  - General Hospital of Thessaloniki ''Hippokratio'', Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital - Hong Kong, Hong Kong
  - Queen Mary Hospital - PPDS, Hong Kong
- Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár, Hungary
- Italy (7):
  - IRCCS Saverio de Bellis-UOSD "Epatopatie", Castellana Grotte
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - ASST Santi Paolo Carlo, S.C. Medicina ad Indirizzo Epatologico e Gastroenterologico, Milan
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale Civile di Baggiovara, Modena
  - A.O.U.P. Paolo Giaccone , U.O.C di Gastroeneterologia, Palermo
  - A.O.U. Pisana, U.O. Epatologia, Pisa
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
- Mexico (6):
  - Clinica de Higado y Gastroenterologia Integral, S.C., Cuernavaca
  - PROACTIVE CR MEXICO SA de CV, Irapuato
  - Consultorio Medico - Distrito Federal, Mexico City
  - Centro De Investigacion Y Gastroenterogia, S.C., México
  - Oaxaca Site Management Organization - Hospital - OSMO - PPDS, Oaxaca City
  - FAICIC, Veracruz
- Poland (2):
  - ID Clinic Arkadiusz Pisula, Mysłowice
  - PlanetMed SP. z. o. o, Wroclaw
- Institutul Clinic Fundeni, Bucharest, Romania
- Changi General Hospital, Singapore, Singapore
- South Korea (10):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Complexo Hospitalario Universitario De Santiago, A Coruña
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron-VIHR, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Switzerland (2):
  - Universitätsspital Bern, Bern
  - Universitätsspital Zürich, Zurich
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan
- Turkey (Türkiye) (10):
  - Adana City Training and Research Hospital, Adana
  - Ankara Bilkent City Hospital, Ankara
  - Gaziantep University Medical Faculty Sahinbey Research and Practice Hospital, Gaziantep
  - Uludag University Medical Faculty, Görükle
  - Ege University, Izmir
  - Katip Celebi University, Karabağlar
  - Kocaeli University Medical Faculty Hospital, Kocaeli
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
  - Marmara University Pendik Training and Research Hospital, Pendik
  - Rize Recep Tayyip Erdogan University Training and Research Hospital, Rize Merkez
- United Kingdom (5):
  - Hull Royal Infirmary, Hull
  - East Suffolk and North Essex NHS Foundation Trust, Ipswich Hospital, Ipswich
  - The Royal London Hospital, London
  - Royal Free Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06051617